CLINICAL TRIAL: NCT07121179
Title: Investigation of Sleep Characteristics in Infants With Joint Hypermobility
Brief Title: Sleep Characteristics in Infants With Joint Hypermobility
Status: Completed | Type: Observational
Sponsor: Nigde Omer Halisdemir University (Other)
Responsible Party: Principal Investigator, Rabia ZORLULAR, principal investigator, Nigde Omer Halisdemir University
Other Study IDs: joint hypermobility
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Joint Hypermobility Syndrome; Sleep; Infant
Keywords: Joint hypermobility; sleep; infant; development
MeSH Terms: conditions — Joint Instability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Joint hypermobility: Joint hypermobility is defined as an increased range of motion in one or more joints compared to the normal range. The Beighton Scoring system is commonly used to distinguish individuals with generalized joint hypermobility from those without. The Beighton Score system includes the following assessments: passive dorsiflexion of the fifth metacarpophalangeal joint, passive hyperextension of the elbow, passive hyperextension of the knee, passive apposition of the thumb to the flexor aspect of the forearm, and forward flexion of the trunk. Infants aged 6-9 months with a Beighton Score > 4 will be included in the joint hypermobility group.
  Interventions: Behavioral: Beighton Scoring system; Behavioral: Brief Infant Sleep Questionnaire
- Healthy infants: A control group consisting of healthy infants, born at term and 6-9-month-old infants without joint hypermobility
  Interventions: Behavioral: Beighton Scoring system; Behavioral: Brief Infant Sleep Questionnaire

INTERVENTIONS:
Behavioral: Beighton Scoring system — The Beighton Scoring system is commonly used to distinguish individuals with generalized joint hypermobility from those without. The Beighton Scoring system includes the following assessments: passive dorsiflexion of the fifth metacarpophalangeal joint, passive hyperextension of the elbow, passive hyperextension of the knee, passive apposition of the thumb to the flexor aspect of the forearm, and forward flexion of the trunk. A Developmental Physiotherapy and Pediatric Rehabilitation specialist will evaluate the joint hypermobility assessment of infants.
Behavioral: Brief Infant Sleep Questionnaire — Infant sleep problems are among the most common problems presented to pediatricians. The extended version of the "Brief Infant Sleep Questionnaire" is a questionnaire developed by Sadeh to assess sleep problems and their causes in early childhood.

SUMMARY:
Joint hypermobility is defined as an increased range of motion in one or more joints compared to the normal range. The Beighton Scoring (BS) system is commonly used to distinguish individuals with generalized joint hypermobility from those without. Passive joint range of motion varies among infants, children, and adults. Since younger children exhibit greater joint mobility than older children and adults, age-specific revisions of the cut-off values are necessary for the diagnosis of Generalized Joint Hypermobility (GJH). To this end, a recent study suggested that children aged 12 to 60 months should be diagnosed with GJH if the BS is greater than 4.

Studies have shown that motor development in children with joint hypermobility is delayed during early childhood, although most children catch up with their peers before the age of two. Infants with joint hypermobility experience significant delays in both gross and fine motor development. Additionally, proprioceptive impairments have been identified in both children and adults with joint hypermobility. A study evaluating sensory processing skills in toddlers with GJH reported sensory processing difficulties compared to their non-GJH peers. A review of the literature reveals that GJH affects the musculoskeletal system, motor development, and sensory processing skills in infants; however, no studies have been found investigating sleep characteristics in infants with GJH. This study aims to investigate the sleep characteristics of term infants aged 6 to 9 months with GJH and to compare them with their non-GJH peers.

DETAILED DESCRIPTION:
Ligamentous laxity and the resulting joint hypermobility are present in various conditions affecting children, such as Marfan syndrome and Ehlers-Danlos syndrome. However, in most cases, joint hypermobility is a limited condition referred to as Generalized Joint Hypermobility (GJH). GJH is defined as asymptomatic hypermobility in more than five joints. The Beighton Scoring (BS) system is commonly used to distinguish individuals with generalized joint hypermobility from those without. The BS system includes the following assessments: passive dorsiflexion of the fifth metacarpophalangeal joint, passive hyperextension of the elbow, passive hyperextension of the knee, passive apposition of the thumb to the flexor aspect of the forearm, and forward flexion of the trunk.

In children older than five years, a cut-off score of ≥6 is used to diagnose GJH. In adults up to 50 years of age, a score of ≥5 out of 9 indicates GJH, while a score of ≥4 out of 9 is considered positive for GJH in adults over 50 years.

Joint hypermobility can cause stability issues in the musculoskeletal system due to connective tissue laxity. This can trigger problems such as discomfort, restlessness, and difficulty finding a position, especially during sleep. Sleep disruptions due to nighttime restlessness or frequent position changes may also occur. Furthermore, most studies on joint hypermobility in the literature primarily involve adults. Early developmental assessments are crucial for preventing developmental delays that may emerge later in life.

ELIGIBILITY:
Inclusion Criteria:

* Term infants
* Infants with joint hypermobility
* Post-term infants between 6 and 9 months old

Exclusion Criteria:

* Premature infants
* Infants with congenital malformations
* Infants diagnosed with metabolic, neurological, or genetic diseases
* Infants with joint hypermobility due to any musculoskeletal disease
* Children whose parents did not volunteer for the study

Ages: 6 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Joint hypermobility is defined as an increased range of motion in one or more joints compared to the normal range.While sleep problems can negatively impact an individual's life at any age, their risk for children with joint hypermobility has not been investigated. Therefore, this study aims to address this gap in the literature by evaluating sleep characteristics in children with Joint hypermobility. Infants aged 6-9 months with a Beighton Score > 4 will be included in the joint hypermobility group.A control group consisting of healthy infants, born at term and 6-9-month-old infants without joint hypermobility
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-08-15 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Brief Infant Sleep Questionnaire | 6 months
  The Brief Infant Sleep Questionnaire (BISQ) will be used to assess sleep. This questionnaire has been translated into Turkish and assesses the sleep environment and sleep problems in infants. It consists of 33 items and is based on parental reports of infant or toddler sleep patterns, which are used to validate the data.The BISQ is a questionnaire that measures the following parameters: Average nighttime sleep duration (hours) Average daytime sleep duration (hours) Average total 24-hour sleep duration (hours) Number of nighttime awakenings Nighttime awake time (minutes) Time it takes to fall asleep Parent perceptions about sleep (e.g., are there any sleep problems?) Comparisons are generally made based on duration and numbers. For example, is the average nightly sleep duration of Group A significantly longer than Group B? Or is the number of nightly awakenings inversely proportional to total sleep duration?

CONTACTS AND LOCATIONS:
Overall Officials: Rabia ZORLULAR, Principal Investigator — Nigde Omer Halisdemir University
Locations (1):
- Nigde Omer Halisdemir University, Niğde, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sedky K, Gaisl T, Bennett DS. Prevalence of Obstructive Sleep Apnea in Joint Hypermobility Syndrome: A Systematic Review and Meta-Analysis. J Clin Sleep Med. 2019 Feb 15;15(2):293-299. doi: 10.5664/jcsm.7636. PMID 30736885
- [Result] Boran, P., et al., Translation into Turkish of the expanded version of the "Brief Infant Sleep Questionnaire" and its application to infants. Marmara Medical Journal, 2014. 27(3): p. 178-183.
- [Result] Sadeh A. A brief screening questionnaire for infant sleep problems: validation and findings for an Internet sample. Pediatrics. 2004 Jun;113(6):e570-7. doi: 10.1542/peds.113.6.e570. PMID 15173539
- [Result] Yildiz A, Yildiz R, Burak M, Zorlular R, Akkaya KU, Elbasan B. An investigation of sensory processing skills in toddlers with joint hypermobility. Early Hum Dev. 2024 May;192:105997. doi: 10.1016/j.earlhumdev.2024.105997. Epub 2024 Apr 2. PMID 38614033